CLINICAL TRIAL: NCT01603082
Title: A Randomized, Open-label Study to Compare the Platelet Inhibition With VerifyNow Assay of Ticagrelor Versus Clopidogrel in Troponin Negative Acute Coronary Syndrome Subjects Undergoing Ad Hoc Percutaneous Coronary Intervention
Brief Title: Ad Hoc Percutaneous Coronary Intervention Study in Acute Coronary Syndrome Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5130L00014
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor - 180 mg loading dose
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel - 600 mg loading dose
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — 180 mg loading dose
  Arms: Ticagrelor
Drug: Clopidogrel — 600 mg loading dose
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to assess the pharmacodynamic effect of ticagrelor in ACS patients undergoing an Ad Hoc PCI

DETAILED DESCRIPTION:
A randomized, open-label, multiple-center, parallel group study to compare the platelet inhibition with VerifyNow assay of ticagrelor versus clopidogrel in troponin negative Acute Coronary Syndrome (ACS) subjects undergoing Ad Hoc percutaneous coronary intervention (PCI)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent before initiation of any study-related procedures
* Male or female patients aged 18 years or older
* Documented acute coronary syndrome and troponin negative and undergoing Ad Hoc percutaneous coronary intervention (PCI)
* Females must be post menopausal or surgically sterile
* Taking aspirin as an anti-platelet medication

Exclusion Criteria:

* Use of any thienopyridine or ticagrelor within 7 days prior to randomization
* Any indication for oral anticoagulant (e.g., atrial fibrillation, mitral stenosis or prosthetic heart valve)
* Contraindication that ticagrelor or clopidogrel should not be administered Patient requires dialysis
* History of intolerance or allergy to aspirin

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn F. Carlson, MD, Study Director — AstraZeneca Pharmaceuticals, Wilmington, DE 19850-5437 USA
Locations (16):
- United States (16):
  - Research Site, Birmingham, Alabama
  - Research Site, San Francisco, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Ypsilanti, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Tupelo, Mississippi
  - Research Site, North Kansas City, Missouri
  - Research Site, Belleville, New Jersey
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tyler, Texas
  - Research Site, Richmond, Virginia

REFERENCES:
- [Derived] Sweeny JM, Angiolillo DJ, Franchi F, Rollini F, Waksman R, Raveendran G, Dangas G, Khan ND, Carlson GF, Zhao Y, Teng R, Mehran R. Impact of Diabetes Mellitus on the Pharmacodynamic Effects of Ticagrelor Versus Clopidogrel in Troponin-Negative Acute Coronary Syndrome Patients Undergoing Ad Hoc Percutaneous Coronary Intervention. J Am Heart Assoc. 2017 Mar 29;6(4):e005650. doi: 10.1161/JAHA.117.005650. PMID 28356282
- [Derived] Angiolillo DJ, Franchi F, Waksman R, Sweeny JM, Raveendran G, Teng R, Zhao Y, Carlson G, Khan N, Mehran R. Effects of Ticagrelor Versus Clopidogrel in Troponin-Negative Patients With Low-Risk ACS Undergoing Ad Hoc PCI. J Am Coll Cardiol. 2016 Feb 16;67(6):603-613. doi: 10.1016/j.jacc.2015.11.044. PMID 26868683

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from 15 actively participating sites in the United States of America, from July 2012 until June 2014.
Pre-assignment Details: Overall, 343 participants were screened; 102 met inclusion/exclusion criteria, 100 were randomized. 96 participants completed treatment and 97 participants completed the study.
Groups:
- Ticagrelor: 180 mg loading dose after diagnostic angiography, followed by 90 mg after 12 hours (± 1 hour), with concomitant acetylysalicylic acid (160 mg to 500mg loading dose followed by a daily maintenance dose of 75 mg to 100 mg)
- Clopidogrel: 600 mg loading dose after diagnostic angiography, with concomitant acetylysalicylic acid (160 mg to 500mg loading dose followed by a daily maintenance dose of 75 mg to 100 mg)
Period: Overall Study
Arm/Group | Ticagrelor | Clopidogrel
Started | 51 (Randomized) | 49 (Randomized)
Completed | 49 (Completed the study.) | 48 (Completed the study)
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Failed inclusion criterion after dosed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set, defined as all participants who signed informed consent, who provided demographic and/or baseline screening assessments, and who were randomized into the study regardless of the participant's randomization and treatment status in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Clopidogrel | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 30 | 66
  >=65 years | 15 | 19 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 34 | 36 | 70
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Black or African American | 11 | 11 | 22
  White | 33 | 33 | 66
  Missing values | 5 | 3 | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 11 | 14 | 25
  Not Reported | 28 | 27 | 55
  Missing values | 7 | 7 | 14
Region of Enrollment [Number; unit: Participants]
  United States | 51 | 49 | 100

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of the P2Y12 Receptor at 2 Hours After Loading Doses of Ticagrelor and Clopidogrel as Measured by P2Y12 Reaction Units (PRU) From VerifyNow™
Description: Participants with low (<150) baseline PRU values were excluded.
Time Frame: 2 hours after the loading dose
Population: Pharmacodynamic (PD) Analysis Set (N=93; 46 on ticagrelor, 47 on clopidogrel) - included all participants with PD data and without a major protocol deviation thought to significantly affect the PD of ticagrelor or clopidogrel. Participants in the PD Analysis Set with low (<150) baseline PRU values were excluded from the analyses.
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 45 | 46
PRU | 98.4 (95.4) | 257.5 (74.5)
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -159.1, 95% CI 2-sided [-194.7 to -123.5], Standard Error of Mean 17.9 — Ticagrelor minus clopidogrel

2. Secondary Outcome: Inhibition of the P2Y12 Receptor at 0.5 Hours, End of PCI, and 8 Hours After Loading Doses of Ticagrelor and Clopidogrel as Measured by PRU From VerifyNow™
Description: Participants with low (<150) baseline PRU values were excluded.
Time Frame: 0.5 hours, end of PCI, and 8 hours after the loading dose
Population: PD Analysis Set. Participants in the PD Analysis Set with low (<150) baseline PRU values were excluded from the analyses.
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 44 | 45
PRU
  0.5 hours | 277.3 (73.8) | 297.7 (69.2)
  8 hours | 43.8 (45.7) | 202.3 (89.1)
  End of PCI (n=41 for ticagrelor) | 264.2 (92.2) | 307.8 (59.5)
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Analysis at 0.5 hours after the loading dose; Test type: Superiority or Other; p = 0.182, t-test, 2 sided; Mean Difference (Final Values) = -20.4, 95% CI 2-sided [-50.5 to 9.7], Standard Error of Mean 15.2 — Ticagrelor minus clopidogrel
Statistical Analysis 2: Comparison: Ticagrelor vs Clopidogrel; Analysis at 8 hours after the loading dose; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -158.5, 95% CI 2-sided [-189.4 to -127.7], Standard Error of Mean 15.5 — Ticagrelor minus clopidogrel
Statistical Analysis 3: Comparison: Ticagrelor vs Clopidogrel; Analysis at end of PCI; Test type: Superiority or Other; p = 0.010, t-test, 2 sided; Mean Difference (Final Values) = -43.6, 95% CI 2-sided [-76.5 to -10.7], Standard Error of Mean 16.5 — Ticagrelor minus clopidogrel

ADVERSE EVENTS:
Time Frame: All adverse events (AEs), including serious AEs were monitored from the point of informed consent through the 14 day follow up period. All vascular events were assessed at each visit and could be reported by participants at any time during the study.
Description: AEs were solicited at each scheduled visit and could be reported by the participant at any time during the study.
Arm/Group | Ticagrelor | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 9/51 | 5/49
Other Adverse Events (participants affected / at risk) | 5/51 | 1/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=51) | Clopidogrel (N=49)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 3 (4)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=51) | Clopidogrel (N=49)
Chest pain (General disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AstraZeneca (AZ) for review at least 60 days in advance of the submission for publication. The Investigators in the Multi-Center (MC) study agree to postpone MC publications until the earlier of the first AZ-authorized publication or up to 18 months from study completion at all sites.